CLINICAL TRIAL: NCT02861716
Title: Intrathecal Dexmedetomidine Versus Fentanyl With Bupivacaine for Postoperative Analgesia in Children Undergoing Major Abdominal Cancer Surgery
Brief Title: Intrathecal Dexmedetomidine Versus Fentanyl With Bupivacaine in Children Undergoing Major Abdominal Cancer Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Rania Mohammed Abd elemam, Director, Clinical Research, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prospective
Record Dates: First submitted 2016-07-29; First posted 2016-08-10 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Intrathecal Dexmedetomidine; Pediatric Cancer Surgery
MeSH Terms: interventions — Bupivacaine; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fentanyl and dexmedetomidine (Experimental): intrathecal bupivacaine (0.5%) 0.4mg/kg plus fentanyl and dexmedetomidine in 2ml volume will be injected slowly over 20 seconds.
  Interventions: Drug: Bupivacaine
- dexmedetomidine and placebo for fentanyl (Active Comparator): intrathecal bupivacaine (0.5%) 0.4mg/kg plus dexmedetomidine 0.2 μg/kg in 2ml volume and placebo (for fentanyl 0.2 μg/kg) it will be injected slowly over 20 seconds.
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine
- fentanyl and placebo for dexmedetomidine (Active Comparator): intrathecal bupivacaine (0.5%) 0.4mg/kg plus fentanyl 0.2 μg/kg in 2ml volume and placebo (for dexmedetomidine 0.2 μg/kg) it will be injected slowly over 20 seconds.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine — premedication with Ondansetron (Zofran®) 0.1 mg/kg and Diazepam ( 0.01 mg/kg ), then general anesthesia will be induced with inhalation of sevoflurane 8% in oxygen via face mask. After that intravenous cannula will be placed, and fluid therapy will be standardized during and after surgery.
  After securing the tube in place, the patients will be placed in the lateral decubitus position and a single dose of intrathecal anesthesia will be performed using a 25 gauge needle (Brown ®, Germany) and free flow of CSF technique. Then children will receive intrathecal bupivacaine (0.5%) 0.4mg/kg body weight in 2ml volume and it will be injected slowly over 20 seconds.
  Other Names: heavy marcaine
Drug: Fentanyl — premedication with Ondansetron (Zofran®) 0.1 mg/kg and Diazepam ( 0.01 mg/kg ), then general anesthesia will be induced with inhalation of sevoflurane 8% in oxygen via face mask. After that intravenous cannula will be placed, and fluid therapy will be standardized during and after surgery.
  After securing the tube in place, the patients will be placed in the lateral decubitus position and a single dose of intrathecal anesthesia will be performed using a 25 gauge needle (Brown ®, Germany) and free flow of CSF technique. Then children will receive intrathecal bupivacaine (0.5%) 0.4mg/kg body weight plus fentanyl 0.2 μg/kg in 2ml volume and it will be injected slowly over 20 seconds.
  Arms: fentanyl and placebo for dexmedetomidine
Drug: Dexmedetomidine — premedication with Ondansetron (Zofran®) 0.1 mg/kg and Diazepam ( 0.01 mg/kg ), then general anesthesia will be induced with inhalation of sevoflurane 8% in oxygen via face mask. After that intravenous cannula will be placed, and fluid therapy will be standardized during and after surgery.
  After securing the tube in place, the patients will be placed in the lateral decubitus position and a single dose of intrathecal anesthesia will be performed using a 25 gauge needle (Brown ®, Germany) and free flow of CSF technique. Then children will receive intrathecal bupivacaine (0.5%) 0.4mg/kg body weight plus dexmedetomidine 0.2 μg/kg in 2ml volume and it will be injected slowly over 20 seconds.
  Other Names: precedex
  Arms: dexmedetomidine and placebo for fentanyl

SUMMARY:
In this study the investigators aim to determine the analgesic effect and side effects of intrathecal fentanyl and dexmedetomidine as adjuvant to local anesthetics in pediatric patients undergoing major abdominal cancer surgeries.

DETAILED DESCRIPTION:
After obtaining approval of the local ethics committee of South Egypt Cancer Institute, Assiut University, Assiut, Egypt, and parent's written informed consent, a randomized double -blinded prospective study will be conducted on (60) pediatric patients.

After applying standard monitors; Pulse oximetry (Spo2), Noninvasive arterial blood pressure, Electrocardiography (ECG), pre-medication with Ondansetron (Zofran®) 0.1 mg/kg and Diazepam (0.01 mg/kg), then general anesthesia will be induced with inhalation of sevoflurane 8% in oxygen via face mask and neuromuscular blockade (atracurium besylate 0.5mg/kg) will be used to facilitate endotracheal intubation. After that an intravenous cannula will be placed, and fluid therapy will be standardized during and after surgery.

After securing the tube in place, patients will be placed in lateral decubitus position and intrathecal anesthesia will be performed using a 25 gauge needle (Brown ®, Germany).

Children will be randomly allocated into 3 groups by using opaque sealed envelopes containing a computer generated randomization schedule. The opaque sealed envelopes are sequentially numbered that will be opened before application of anesthetic plan and each group will include (20) patients:

Group (1): children will receive intrathecal bupivacaine (0.5%) 0.4mg/kg in 2ml volume; it will be injected slowly.

Group (2): children will receive intrathecal bupivacaine (0.5%) 0.4mg/kg plus fentanyl 0.2 μg/kg in 2ml volume; it will be injected slowly.

Group (3): children will receive intrathecal bupivacaine (0.5%) 0.4mg/kg plus dexmedetomidine 0.2 μg/kg in 2ml volume; it will be injected slowly.

Anesthesia will be maintained with oxygen, sevoflurane, atracurium besylate (0.15mg/kg) as muscle relaxant and controlled mechanical ventilation. The inhaled concentration of sevoflurane will be adjusted to achieve hemodynamic changes< 30% of the baseline values. No other narcotics, analgesics or sedatives will be administrated intra-operatively.

During surgery, children will receive lactated ringer's solution 6ml/kg/hr, whereas dextrose 50mg/ml in Nacl 4.5mg/ml will be infused at 4ml/kg/hr in the postoperative period.

Heart rate (HR), noninvasive arterial blood pressure (systolic, and diastolic), oxygen saturation (Spo2) will be recorded at baseline (pre-operatively) and every 10 minutes intra-operative till the end of the operation. The occurrence of intra-operative hypo-tension requiring a fluid bolus, and bradycardia requiring atropine will be recorded.

At the end of the surgery, the residual neuromuscular blocking will be reversed using a mixture of atropine (0.02mg/kg) and neostigmine (0.05mg/kg).

Then after extubation, patients will be transmitted to the post anesthesia care unit (PA CU), and will be followed up by:

* Vital signs (heart rate, noninvasive arterial blood pressure, oxygen saturation and respiratory rate) immediately postoperative (0 hour) and at 2, 4, 6, 8, 12,18 and 24 hours of the postoperative period.
* The face, Legs, Activity, Crying, and Consolability (FLACC) pain score with its 0- 10 score range will be used to assess pain immediately postoperative and at 2, 4, 6, 12, 18, 24 hours postoperative.
* The time of first request for analgesia (Intravenous paracetamol 20mg/kg (perfalgan ®) which will be given when the FLA CC score ≥4 and total paracetamol consumption also will be recorded in the 24 hours postoperative.
* The level of sedation will be recorded using Ramsey sedation scale as the same time points of FLA CC score.
* Postoperative adverse effects such as nausea, vomiting, itching, hypo-tension, bradycardia, arrhythmia and respiratory depression (respiratory depression will be defined as decreased Spo2of less than 95% or respiratory rate less than 10 per minute) will be treated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* Patients scheduled for major abdominal cancer surgeries, expected to last more than 90 minutes

Exclusion Criteria:

* Sacral bone abnormalities
* Spina bifida
* Coagulopathy
* Mental delay or retardation
* Known allergy to the study drugs
* Local infection at the site of injection

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-02 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain by Face, Legs, Activity, Crying, and Consolability (FLACC) Pain Score | one day
  FLA CC pain score will be assessed immediately postoperative and then every 2 hours. Each item is scored 0 to 2, yielding a total between 0 and10

SECONDARY OUTCOMES:
Recurrence of pain | 24 hours
  return of any pain during the specified post-dose period

CONTACTS AND LOCATIONS:
Overall Officials: rania abdelemam, lecturer, Principal Investigator — South Egypt Cancer Institute
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcome measures will be made available within 6 months of study completion